CLINICAL TRIAL: NCT03525964
Title: Individualized Treatment for Acute Achilles Tendon Rupture Based on Barfod's Ultrasonographic Length Measure - a Randomized Controlled Trial
Brief Title: Individualized Treatment of Acute Achilles Tendon Rupture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Jutland Regional Hospital (Other)
Collaborators: The Danish Rheumatism Association (Other)
Responsible Party: Principal Investigator, Marianne Toft Vestermark, Head of Orthopaedic Resaerch, MD PhD, Central Jutland Regional Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Viborg NVK 1-10-72-428-17
Record Dates: First submitted 2018-03-20; First posted 2018-05-16 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Achilles Tendon Rupture
Keywords: Individualized treatment; Functional outcome

STUDY DESIGN:
Intervention Model Description: Prospective
Who Masked: Investigator, Outcomes Assessor
Masking Description: The posterior site of the achilles tendon region is covered by dark tape during the functional assesments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Individualized treatment (Experimental): The ruptured achilles tendon is examined by ultrasonography. If the overlap of the tendon ends is less than 25 % or the tendon is elongated 7 % or more the patient receives conventional open operative treatment. The tendon is sutured with double fiberwire size 2 a.m. Kessler under prophylactic Dicloxacillin 2 g and in local anaesthesia or alternatively popliteal or spinal block. The injured leg is placed in a circulated below-the-knee cast after surgery. The ankle is held at maximal, unforced plantar flexion. Weight bearing is not allowed and the patient should walk with the aid of crutches. After 3 weeks from initiated treatment in the Emergency Department the cast is removed in the Outpatients Department and the injured leg is transferred to a functional brace (Walker boot) with 3 heel wedges promoting 20 degrees plantar flexion over the ankle.
  The patient will follow standard functional rehabilitation and the follow-up evaluations.
  Interventions: Procedure: Individualized treatment of Acute Achilles tendon rupture.
- Control group 1 (Active Comparator): For the patients allocated to non-operative treatment the injured leg is placed in a circulated below-the-knee cast from the time of the first appointment in the Outpatients Department. The ankle is held at maximal, unforced plantar flexion. Weight bearing is not allowed and the patient should walk with the aid of crutches. After 3 weeks from initiated treatment in the Emergency Department the cast is removed in the Outpatients Department and the injured leg is transferred to a functional brace (Walker boot) with 3 heel wedges promoting 20 degrees plantar flexion over the ankle.
  The patient will follow standard functional rehabilitation and the follow-up evaluations.
  Interventions: Procedure: Non-operative treatment
- Control group 2 (Active Comparator): The tendon is sutured with double fiberwire size 2 a.m. Kessler under prophylactic Dicloxacillin 2 g and in local anaesthesia or alternatively popliteal or spinal block. The injured leg is placed in a circulated below-the-knee cast from the time of the first appointment in the Outpatients Department. The ankle is held at maximal, unforced plantar flexion. Weight bearing is not allowed and the patient should walk with the aid of crutches. After 3 weeks from initiated treatment in the Emergency Department the cast is removed in the Outpatients Department and the injured leg is transferred to a functional brace (Walker boot) with 3 heel wedges promoting 20 degrees plantar flexion over the ankle.
  The patient will follow standard functional rehabilitation and the follow-up evaluations.
  Interventions: Procedure: Operative treatment

INTERVENTIONS:
Procedure: Individualized treatment of Acute Achilles tendon rupture. — The most proximal border of the calcaneus and the most distal point of the musculotendinous junction of the Achilles tendon and the medial gastrocnemius muscle is identified and marked on the skin. These two points on the un-injured leg defines the original length of the total Achilles tendon and consist of the free tendon and the fascia [1]. The difference in length between the injure and the un-injured leg determines elongation for the ruptured Achilles tendon. The relative elongation of the ruptured tendon together with overlap of the tendon ends on the cross-sectional area determines the treatment for the patients receiving individualized treatment: 1) patients with 0-6% elongation of the tendon and a minimum of 25% tendon are treated non-operatively 2) patients with 7% elongation or more or less than 25% tendon overlap are treated operatively. The cut-off at 7% elongation is determined for 75% sensitivity and 65% specificity of elongation.
  Arms: Individualized treatment
Procedure: Non-operative treatment — Circulated cast below the knee in maximal, unforced plantar flexion over the ankel.
  Arms: Control group 1
Procedure: Operative treatment — Open surgery with suture of the ruptured achilles tendon prior to circulated cast below the knee in maximal, unforced plantar flexion over the ankel.
  Arms: Control group 2

SUMMARY:
To asses the functional outcome after individualized treatment of acute achilles tendon rupture. The treatment is individualizes on the basis of ultrasonographic status of tendon overlap and Barfod's Ultrasonographic length measure. Patients are allocated for operative treatment if there the tendon overlap is less than 25 % or the tendon is elongated with 7% or more compared to the healthy, contralateral achilles tendon.

The study includes two control groups of non-operative and operative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Appointment in the Outpatients Department within 4 days of injury.
* Total Achilles tendon rupture.
* Initial treatment with split cast with the ankle in maximal plantar flexion must be started within 24 hours of injury.
* The patient must be expected to be able to attend rehabilitation and post-examinations.
* The patient must be able to speak and understand Danish.
* The patient must be able to give informed consent.

Exclusion Criteria:

* Rupture of the Achilles tendon either at the insertion on the calcaneus or at musculotendinous junction of the triceps surae.
* Previous rupture of the Achilles tendon in any of the two legs.
* Treated with Fluoroquinolones or corticosteroids within the last 6 months.
* In medical treatment of diabetes.
* Suffers from rheumatic disease.
* Other conditions prior to the injury resulting in reduced function of any of the two legs.
* Contra-indication for surgery: severe arthrosclerosis with no palpable pulse in the foot, broken skin in the Achilles region of the injured leg.
* Inability to lie in prone position on the operating table.
* Terminal illness or severe medical illness: ASA (American Society of Anesthesiologists) score higher than or equal to 3.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Heel-rise work test | Evaluation method after 12 months of started treatment
  An endurance test where the patient stands on one leg and lifts the heel up and down until exhaustion. The number and the height of the heel rises are counted and measured and plotted into a diagram on an X-axis and Y-axis respectively. The results are then compared to the weight of the patient and the total work is estimated as area under the curve. The heel lift distance between the heel and the floor is measured in millimeters. The procedure is performed on the uninjured leg first and subsequently on the injured leg. The patient is barefoot for the heel-rise work test and stands on a flat surface with a 10 degree inclination.
  For these functional tests a measurement system MuscleLab (Ergotest Technology, Oslo, Norway) will be used at all the centers.

SECONDARY OUTCOMES:
Barfod's ultrasonographic length measure | Evaluation method after 6 and 12 months of started treatment
  The examination of both the total and the free part of the achilles tendon of both the injured and un-injured leg is performed. The total length of the tendon is defined under the description of the intervention. The free part of the achilles tendon is defined as the distance between the proximal border of calcaneus and the musculotendinous junction of the soleus muscle and the achilles tendon. The method will be used both diagnostically for the individualized treatment and as a secondary endpoint.
Indirectly, clinical Achilles tendon length estimate | Evaluation method after 6 and 12 months of started treatment
  Achilles tendon length is indirectly estimated clinically by use of the Achilles Tendon Resting Angle (ATRA) or the Achilles Tendon Length Measure (ATLM). The patient lies flat in prone position on the examination bed. The knee is flexed at 90 degrees and the ankle sits in relaxed position. The ATRA is determined as the angle between the corpus of the fibula and the corpus of the 5th metatarsus. The ATLM is determined as the distance from the caput of the 5th metatarsus to the surface of the examination bed. Both the ATRA and the ATLM are determined for both the injured and the uninjured leg. The difference between the healthy and the injured leg is evaluated
Complications | Evaluation method after 12 months of started treatment
  Incidence rate of the commonly known complications and adverse events such as infection, re-rupture, permanent sural nerve dysfunction, adhesions and pain at the scar is noted. Attention is also paid to so far unknown complications in relation to the treatments.
Achilles tendon Total Rupture Score (ATRS) | Evaluation method after 6 and 12 months of started treatment
  Patients will fill out the ATRS questionnaire in connection to the follow-up visits in the Outpatients Department. ATRS is a patient-reported outcome measure.
  This questionnaire is a part of the usual examination of the patients' function, and is used during all follow-ups in the usual care.
Heel-rise Work test | Evaluation method after 6 months of started treatment
  An endurance test where the patient stands on one leg and lifts the heel up and down until exhaustion. The number and the height of the heel rises are counted and measured and plotted into a diagram on an X-axis and Y-axis respectively. The results are then compared to the weight of the patient and the total work is estimated as area under the curve. The heel lift distance between the heel and the floor is measured in millimeters. The procedure is performed on the uninjured leg first and subsequently on the injured leg. The patient is barefoot for the heel-rise work test and stands on a flat surface with a 10 degree inclination.
  For these functional tests a measurement system MuscleLab (Ergotest Technology, Oslo, Norway) will be used at all the centers.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne T Vestermark, MD PhD, Principal Investigator — Central Jutland Regional Hospital
Locations (4):
- Denmark (4):
  - Copenhagen University Hospital, Hvidovre, Hvidovre
  - Hospital Lillte Belt, Kolding, Kolding
  - Zealand University Hospital, Køge, Køge
  - Jutland Central Regional Hospital, Viborg

IPD SHARING:
Plan to Share IPD: No
There is no plan of sharing data with researchers not already included in this study.

REFERENCES:
- [Background] Barfod KW, Riecke AF, Boesen A, Hansen P, Maier JF, Dossing S, Troelsen A. Validation of a novel ultrasound measurement of achilles tendon length. Knee Surg Sports Traumatol Arthrosc. 2015 Nov;23(11):3398-406. doi: 10.1007/s00167-014-3175-2. Epub 2014 Jul 20. PMID 25038882
- [Derived] Hansen MS, Vestermark MT, Holmich P, Kristensen MT, Barfod KW. Individualized treatment for acute Achilles tendon rupture based on the Copenhagen Achilles Rupture Treatment Algorithm (CARTA): a study protocol for a multicenter randomized controlled trial. Trials. 2020 May 12;21(1):399. doi: 10.1186/s13063-020-04332-z. PMID 32398120